CLINICAL TRIAL: NCT02183012
Title: Open-label, Randomised, Single Dose, Four-way Crossover Study to Investigate the Relative Bioavailability of a 400 mg Ibuprofen Extrudate Tablet Compared to a 400 mg Ibuprofen Lysinate Tablet (Dolormin Extra®) and a 400 mg Ibuprofen Tablet (Brufen® 400 mg, Denmark) in Fasted Condition and After Ingestion of a Standardised Meal in Healthy Male and Female Volunteers.
Brief Title: Study to Investigate the Relative Bioavailability of Ibuprofen in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1024.5
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — solufenum; Ibuprofen

ARMS (6):
- A: Ibuprofen extrudate, fed state (Experimental)
  Interventions: Drug: Ibuprofen extrudate
- B: Ibuprofen extrudate, fasted state (Experimental)
  Interventions: Drug: Ibuprofen extrudate
- C: Ibuprofen lysinate tablet, fed state (Active Comparator)
  Interventions: Drug: Ibuprofen lysinate
- D: Ibuprofen lysinate tablet, fasted state (Active Comparator)
  Interventions: Drug: Ibuprofen lysinate
- E: Ibuprofen tablet, fed state (Active Comparator)
  Interventions: Drug: Ibuprofen
- F: Ibuprofen tablet, fasted state (Active Comparator)
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen extrudate
  Arms: A: Ibuprofen extrudate, fed state; B: Ibuprofen extrudate, fasted state
Drug: Ibuprofen lysinate
  Arms: C: Ibuprofen lysinate tablet, fed state; D: Ibuprofen lysinate tablet, fasted state
Drug: Ibuprofen
  Arms: E: Ibuprofen tablet, fed state; F: Ibuprofen tablet, fasted state

SUMMARY:
* Study to demonstrate average bioequivalence between a 400 mg ibuprofen extrudate tablet (Test) and a 400 mg ibuprofen lysinate tablet (Dolormin extra ®; reference 1) under fasted conditions.
* Study to determine the relative bioavailability of ibuprofen following single administration of a 400 mg ibuprofen extrudate tablet (Test) compared to a 400 mg ibuprofen tablet (Brufen® 400mg, Denmark; Reference 2) under fasted conditions.
* Study to determine the relative bioavailability of ibuprofen following single administration of a 400 mg ibuprofen extrudate tablet (Test) compared to a 400 mg ibuprofen lysinate tablet (Dolormin extra ®; reference 1) or a 400 mg ibuprofen tablet (Brufen® 400mg, Denmark; Reference 2), respectively, under fed conditions.
* Study to evaluate the effect of food on the pharmacokinetics of ibuprofen for all three formulations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females according to the following criteria:

  * Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests:

    * No finding deviating from normal and of clinical relevance
    * No evidence of a clinically relevant concomitant disease.
* Age ≥ 21 and Age ≤ 50 years
* BMI ≥ 18.5 and BMI ≤ 29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP (Good Clinical Practice) and the local legislation

Exclusion Criteria:

* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* History of recent surgery including dental surgery
* History of gastrointestinal ulcer or gastrointestinal inflammation (gastritis, ulcerative colitis, Crohn's disease)
* Blood dyscrasias of unknown origin
* Subjects with porphyries diseases
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity/allergic rhinitis (including drug allergy) which is deemed relevant to he trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial except substitution therapy (thyroid, ovaries) and hormonal contraception
* Use of any drugs, which might influence the results of the trial (within 10 days prior to administration or during the trial)
* Participation in another trial with an investigational drug (within two months prior to administration or during the trial)
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range of clinical relevance
* Inability to comply with dietary regimen of study centre
* For female subjects:

  * Pregnancy
  * Positive pregnancy test
  * No adequate contraception e.g. oral contraceptives, sterilisation, IUP (intrauterine pessary: in case a IUP was used for contraception, volunteers must be advised to employ additional contraceptive measures (e.g. condom by partner) because prostaglandin inhibition may alter IUP contraceptive efficacy)
  * Inability to maintain this adequate contraception during the whole study period
  * Lactation period

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2002-08; Primary Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma from zero time to infinity) | Pre-dose and 15, 30, 45 min, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24 hours after treatment on day 1 of visits 2-5
Cmax (maximum observed concentration of the analyte in plasma) | Pre-dose and 15, 30, 45 min, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24 hours after treatment on day 1 of visits 2-5
AUC0-tz (area under the concentration-time curve of the analyte in plasma from zero time to the time of the last quantifiable drug concentration) | Pre-dose and 15, 30, 45 min, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24 hours after treatment on day 1 of visits 2-5

SECONDARY OUTCOMES:
Individual time courses of the ibuprofen plasma concentrations | Pre-dose and 15, 30, 45 min, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24 hours after treatment on day 1 of visits 2-5
AUCtrunc (Area under the concentration-time curve of the analyte in plasma from zero time to median tmax values of the reference formulation) | Pre-dose and 15, 30, 45 min, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24 hours after treatment on day 1 of visits 2-5
tmax (time to reach Cmax) | Pre-dose and 15, 30, 45 min, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24 hours after treatment on day 1 of visits 2-5
t1/2 (terminal half-life of the analyte in plasma) | Pre-dose and 15, 30, 45 min, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24 hours after treatment on day 1 of visits 2-5
λz (terminal rate constant of the analyte in plasma) | Pre-dose and 15, 30, 45 min, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24 hours after treatment on day 1 of visits 2-5
MRTtot (total mean residence time of the analyte molecules in the body) | Pre-dose and 15, 30, 45 min, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24 hours after treatment on day 1 of visits 2-5
CL/F (total clearance of the analyte in plasma following extravascular administration) | Pre-dose and 15, 30, 45 min, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24 hours after treatment on day 1 of visits 2-5
Vz/F (apparent volume of distribution during the terminal phase λz following extravascular administration) | Pre-dose and 15, 30, 45 min, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24 hours after treatment on day 1 of visits 2-5
Number of patients with adverse events | up to 24 days
Number of patients with abnormal changes in laboratory parameters | up to 8 days following last drug administration
Number of patients with clinically significant changes in vital signs (blood pressure (BP), pulse rate (PR)) | up to 8 days following last drug administration
Number of patients with abnormal changes in 12-lead electrocardiogram (ECG) | up to 8 days following last drug administration
Number of patients with abnormal findings in physical examination | up to 8 days following last drug administration
Assessment of tolerability on a 4-point scale | up to 8 days following last drug administration